CLINICAL TRIAL: NCT00624598
Title: Phase I Study of Integrating RMR Technology and Email Counseling in a PCP Office.
Brief Title: The Short-Term Effect of a Technology Driven Weight Control (SMART) Program for Obese Adults
Acronym: WCPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado Center for Chronic Care Innovations, Inc. (Other)
Collaborators: Microlife (Industry)
Responsible Party: Scott McDoniel, Capella University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C41 # 001
Record Dates: First submitted 2008-02-19; First posted 2008-02-27 (Estimated); Last update posted 2008-09-17 (Estimated); Status verified 2008-09

CONDITIONS: Obesity; Hypertension
MeSH Terms: conditions — Obesity; Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMART Group (Experimental): The experimental group will have a nutrition program based solely on measured resting metabolic rate. The nutrition plan will be a specific calorie level that will promote a 1-2.5 lb per week weight reduction. No experimental participants' nutrition plan will be below 1200 Kcal/day for women or 1600 Kcal/day for men. Second, the experimental group will receive a downloadable copy of a computerized nutrition software program (BalanceLog: Microlife USA, Inc. Golden, CO) that functions s on a Windows 2000-XP or Palm operating system.
  Interventions: Behavioral: SMART
- Usual Care (Active Comparator): Standard 1200 kcal/day diet (women) 1600 kcal/day diet (men) using a sample 3-day menu program. The diet will be follow current government based recommendations for carbohydrates (i.e. 55%), fat (30%), and protein (15%). Study participants will receive a standard paper-based food and exercise journal
  Interventions: Behavioral: SMART

INTERVENTIONS:
Behavioral: SMART — Use of measured resting metabolic rate from indirect calorimetry for personalized diet program and use of a computer application for journalizing food and exercise.

SUMMARY:
The purpose of this study is to evaluate the short-term effect of a technology based weight reduction program for obese (BMI > 30 kg/m2) adults in a primary care office.

ELIGIBILITY:
Inclusion Criteria:

1. Participant between the ages of 18-65 years.
2. Participant with a BMI (Body Mass Index > 30.0 kg/m2)
3. Have access and use email a minimum of 2-days per week.

Exclusion Criteria:

1. Participant is not pregnant or lactating: Weight loss is not recommended for pregnant women and extra energy requirements are essential for fetal development (Butte, Wong, Treuth, Ellis, & O'Brian Smith, 2004; Durnin, 1991).
2. Participant is not currently participating in any structured/self-help weight loss program. The elimination of individuals actively participating in a current weight loss program will reduce the potential of a carry-over effect from these weight loss modalities (Fife-Shaw, 2006).
3. Participant has not attempted weight loss in the past 3 months. Same as number two.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Individuals receiving a technology-based weight reduction program will not have a significant increase in psychosocial constructs (i.e. weight self-efficacy, perceived behavioral control, attitude) compared to control group. | 10 weeks
Individuals receiving a technology-based weight reduction program will not improve eating behaviors (i.e. dietary cognitive restraint, emotional eating, uncontrolled eating) compared to control group. | 10 weeks
Individuals receiving a technology-based weight reduction program will not lose significantly more weight compared to control group. | 10 weeks
Individuals receiving a technology-based weight reduction program will not significantly improve systolic and diastolic blood pressure compared to control group(controlled for Bp medications). | 10 Weeks

SECONDARY OUTCOMES:
Individuals receiving a technology-based weight reduction program will not significantly improve weight quality of life compared to control group. | 10 weeks
There is no relationship between psychosocial values (i.e. weight self-efficacy, weight perceived behavioral control, weight attitude) and eating behaviors (i.e. dietary cognitive restraint, uncontrolled eating, and emotional eating). | 10 Weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Westmed Family Healthcare, Westminster, Colorado
  - Westminster Medical Center, Westminster, Colorado